CLINICAL TRIAL: NCT06613789
Title: A Partially Randomized Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of 426c.Mod.Core-C4b Vaccine Adjuvanted With 3M-052-AF + Alum in Infants With Perinatal HIV Exposure Who Are Without HIV at Birth
Brief Title: Safety & Immunogenicity of 426c.Mod.Core-C4b Vaccine With 3M-052-AF+Alum in Infants Perinatally Exposed to HIV But Uninfected
Acronym: HVTN316
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Fred Hutchinson Cancer Center (Other); Access to Advanced Health Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 316; UM1AI068614 (NIH)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: HIV
MeSH Terms: conditions — HIV Infections | interventions — aluminum sulfate

STUDY DESIGN:
Intervention Model Description: Part A is dose escalating. Part B is parallel.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Part A, Group 1: 426c.Mod.Core-C4b (20 mcg) (Experimental): Participants will receive 426c.Mod.Core-C4b (20 mcg) alone to be administered as two 0.25-mL intramuscular (IM) doses, one into each thigh at weeks 0, 12, and 28.
  Interventions: Biological: 426c.Mod.Core-C4b
- Part A, Group 2: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (0.3 mcg) + Alum (250 mcg) (Experimental): Participants will receive 426c.Mod.Core-C4b (20 mcg) admixed with 3M-052-AF (0.3 mcg) and aluminum hydroxide suspension (Alum) (250 mcg) to be administered as two 0.25-mL IM doses, one into each thigh at weeks 0, 12, and 28.
  Interventions: Biological: 426c.Mod.Core-C4b; Biological: 3M-052-AF; Biological: Aluminum hydroxide suspension (Alum)
- Part A, Group 3: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (0.75 mcg) + Alum (250 mcg) (Experimental): Participants will receive 426c.Mod.Core-C4b (20 mcg) admixed with 3M-052-AF (0.75 mcg) and aluminum hydroxide suspension (Alum) (250 mcg) to be administered as two 0.25-mL IM doses, one into each thigh at weeks 0, 12, and 28.
  Interventions: Biological: 426c.Mod.Core-C4b; Biological: 3M-052-AF; Biological: Aluminum hydroxide suspension (Alum)
- Part A, Group 4: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (1.5 mcg) + Alum (250 mcg) (Experimental): Participants will receive 426c.Mod.Core-C4b (20 mcg) admixed with 3M-052-AF (1.5 mcg) and aluminum hydroxide suspension (Alum) (250 mcg) to be administered as two 0.25-mL IM doses, one into each thigh at weeks 0, 12, and 28.
  Interventions: Biological: 426c.Mod.Core-C4b; Biological: 3M-052-AF; Biological: Aluminum hydroxide suspension (Alum)
- Part B, Group 5: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (TBD)* + Alum (250 mcg) (Active Comparator): Participants will receive 426c.Mod.Core-C4b (20 mcg) admixed with 3M-052-AF (TBD) and Alum (250 mcg) to be administered as two 0.25-mL IM doses, one into each thigh at weeks 0, 12, and 28.
  Interventions: Biological: 426c.Mod.Core-C4b; Biological: 3M-052-AF; Biological: Aluminum hydroxide suspension (Alum)
- Part B, Group 6: Placebo (Placebo Comparator): Participants will receive Placebo (Tris Sodium Chloride (NaCl) buffer ) to be administered as two 0.25-mL IM doses, one into each thigh at weeks 0, 12, and 28.
  Interventions: Biological: Placebo and Diluent

INTERVENTIONS:
Biological: 426c.Mod.Core-C4b — self-assembling nanoparticle expressing up to 7 molecules of the 426c.Mod.Core envelope immunogen.
  Arms: Part A, Group 1: 426c.Mod.Core-C4b (20 mcg); Part A, Group 2: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (0.3 mcg) + Alum (250 mcg); Part A, Group 3: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (0.75 mcg) + Alum (250 mcg); Part A, Group 4: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (1.5 mcg) + Alum (250 mcg); Part B, Group 5: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (TBD)* + Alum (250 mcg)
Biological: 3M-052-AF — 3M-052-AF is an aqueous formulation (AF) of a lipidated small molecule imidazoquinoline that is a Toll-like receptor (TLR)7/8 and inflammasome agonist. To be administered as 0.3 mcg, 0.75 mcg, or 1.5 mcg admixed with 426c.Mod.Core-C4b, with Alum
  Arms: Part A, Group 2: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (0.3 mcg) + Alum (250 mcg); Part A, Group 3: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (0.75 mcg) + Alum (250 mcg); Part A, Group 4: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (1.5 mcg) + Alum (250 mcg); Part B, Group 5: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (TBD)* + Alum (250 mcg)
Biological: Aluminum hydroxide suspension (Alum) — Aluminum hydroxide suspension (Alum) to be administered as 250 mcg (aluminum content) admixed with 426c.Mod.Core-C4b with 3M-052-AF.
  Arms: Part A, Group 2: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (0.3 mcg) + Alum (250 mcg); Part A, Group 3: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (0.75 mcg) + Alum (250 mcg); Part A, Group 4: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (1.5 mcg) + Alum (250 mcg); Part B, Group 5: 426c.Mod.Core-C4b (20 mcg) + 3M-052-AF (TBD)* + Alum (250 mcg)
Biological: Placebo and Diluent — Tris-NaCl buffer.
  Arms: Part B, Group 6: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of 426c.Mod.Core-C4b vaccine adjuvanted with 3M-052-AF + Alum in infants with perinatal HIV exposure who are without HIV at birth

DETAILED DESCRIPTION:
This study will compare the safety and immunogenicity of an experimental HIV vaccine in infants with perinatal HIV exposure who are without HIV at birth. The study vaccine is called 426c.Mod.Core-C4b. The vaccine is mixed with an adjuvant called 3M-052-AF + Alum.

This study is divided into 2 parts: Part A and B. Part A has 4 groups, while Part B has 2 groups. Part A of the study is testing the vaccine alone or in combination with different doses of adjuvant. Part B is testing study vaccine and the safest dose of adjuvants from Part A versus placebo. Depending on their group, participants will receive 426c.Mod.Core-C4b, 426c.Mod.Core-C4b vaccine adjuvanted with 3M-052-AF + Alum, or a placebo by injection at Months 0, 3, and 7.

Additional study visits will occur at Day 1, Week 2, Month 3 1/2, Month 7 1/2, Month 10, Year 1, Year 1 1/2, and Year 1 3/4. Study visits may include physical exams, blood and saliva collection for the infants and questionnaires, counselling, blood, and optional breastmilk collection for the mothers of infants.

ELIGIBILITY:
Inclusion Criteria: Mother

* Mother's age is at least 18 years and is willing and able to provide written informed consent for their and their infant's participation in this study
* Mother is in the second or third trimester of singleton pregnancy, as determined by a clinical exam or sonography and reported menstrual history
* Mother agrees to donate umbilical cord blood
* Mother has a planned Caesarian delivery at Chris Hani Baragwanath Academic Hospital (Soweto) and plans to remain in the area after delivery and through study duration
* Mother is determined by the site investigator to be in good overall health at the time of delivery based on medical history and physical exam
* Mother has a documented CD4 count of more than 350 cells/mcL at screening
* Mother has been on cART for at least 16 weeks prior to delivery and intends to continue with cART for the duration of breastfeeding
* Mother has a viral load of less than 400 copies/mL between 2 weeks before and 7 days after delivery
* Mother has access to the participating HVTN CRS and is willing to be followed for the planned duration of the study
* Mother demonstrates understanding of this study and is able and willing to complete the informed consent process and delivery with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Mother agrees not to enroll either self or infant in another research study for the duration of the trial without prior approval of the HVTN 316 PSRT.
* Mother has confirmed positive HIV-1 status documented by medical records at any time during or prior to screening, and confirmed by the HVTN CRS by serology

Exclusion Criteria: Mother

* Any World Health Organization (WHO) grade IV illness within 1 year prior to study enrollment, as determined by the history and physical examination and review of the medical record (if available). These include HIV wasting syndrome; PJP pneumonia; cerebral toxoplasmosis; extrapulmonary cryptococcosis; progressive multifocal leukoencephalopathy; any disseminated endemic mycosis (histoplasmosis); candidiasis of the esophagus, trachea, bronchi, or lung; disseminated atypical mycobacteria; non-typhoid salmonella septicemia; extrapulmonary tuberculosis; lymphoma; and Kaposi's sarcoma.
* Prior participation in any HIV-1 vaccine or anti-HIV antibody-mediated prevention trial
* Receipt of any investigational agent during this pregnancy
* Receipt of blood products, immunoglobulin (Ig), or immunomodulating therapy within 45 days prior to, and the day of delivery
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of infant safety or reactogenicity, or a volunteer's ability to give informed consent
* Any condition that places the newborn at higher risk of early-onset sepsis, such as concern for active maternal infection at delivery, as determined by local site investigators (eg, fever)
* Detectable hepatitis B surface antigen (HBsAg)

Inclusion Criteria: Infant

* Born via Caesarean delivery to a pregnant woman living with HIV-1 who meets all maternal inclusion/exclusion criteria listed above
* Estimated gestational age at birth is at least 37 weeks

Note: If gestational age at birth is not documented in the infant's available birth records, study staff may assess gestational age at the earliest possible opportunity during the screening period and use this assessment for purposes of eligibility determination.

* Weight at birth is at least 2.5 kg
* Has initiated ARV prophylaxis consistent with current site-specific standard of care
* Hemoglobin (HgB) more than 14.0 g/dL
* White blood cell (WBC) count ≥ 7,000 cells/mm3
* Platelets more than 100,000 cells/mm3
* Alanine aminotransferase (ALT) less than 1.25 times upper limit of age-adjusted normal
* Creatinine less than 1.1 times upper limit of age adjusted normal
* Negative HIV-1 nucleic acid test (NAT) on specimen drawn within 72 hours of birth
* Written informed consent provided by mother
* Age is equal to or less than 7 days

Exclusion Criteria: Infant

* Any clinically significant congenital anomaly/birth defect
* Documented or suspected serious medical illness, infection, clinically significant finding from physical examination, or immediate life-threatening condition, including requirement for ongoing supplemental oxygen, as judged by the examining clinician
* Receipt of or anticipated need for blood products, immunoglobulin, or immunosuppressive therapy. This includes infants who require hepatitis B immunoglobulin (HBIG), but it does not require exclusion of infants who receive hepatitis B vaccine in the newborn period.
* Receipt of any other investigational product

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2026-07-13 (Estimated); Primary Completion 2027-06-03 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting local reactogenicity signs and symptoms and number of local reactogenicity signs and symptoms experienced by each participant | Measured through 14 days following receipt of study product at day 5, week 12, and week 28
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Number of participants reporting systemic reactogenicity signs and symptoms symptoms and number of systemic reactogenicity signs and symptoms experienced by each participant, | Measured through 14 days following receipt of study product at day 5, week 12, and week 28
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Number of participants reporting adverse events and overall number of adverse events | Measured through out the study period
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Number of participants reporting serious adverse events and overall number of serious adverse events | Measured through 12 months post last vaccination at week 28
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Number of participants reporting medically attended adverse events and overall number of medically attended adverse events | Measured through 12 months post last vaccination at week 28
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Number of participants reporting adverse events of special interest (AESIs) that are Potential Immune Mediated Medical Conditions (PIMMCs) and overall number of AESIs that are PIMMCs | Measured through 12 months post last vaccination at week 28
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Number of participants reporting AEs leading to early participant withdrawal or permanent discontinuation | Measured through 12 months post last vaccination at week 28
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [March 2017]
Response rate of CD4bs-specific IgG binding antibodies | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by binding antibody multiplex assay (BAMA)
Magnitude of CD4bs-specific IgG binding antibodies | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by binding antibody multiplex assay (BAMA)
Response rate of CD4bs-specific memory B cells | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by flow cytometry
Magnitude of CD4bs-specific memory B cells | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by flow cytometry

SECONDARY OUTCOMES:
Response rate of serum Ab neutralization of vaccine-matched viruses | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by TZM-bl pseudoneutralization assay
Magnitude of serum Ab neutralization of vaccine-matched viruses | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by TZM-bl pseudoneutralization assay
Differential neutralization of HIV-1 strains that are diagnostic for CD4bs bNAb precursors | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by TZM-bl assay
Response rate of serum Ab neutralization of heterologous HIV-1 strains | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by TZM-bl assay
Magnitude of serum Ab neutralization of heterologous HIV-1 strains | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by TZM-bl assay
Response rate (i.e., percentage) of CD4bs-specific, including VRC01-class, B cells | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by BCR sequencing of sorted B cells
Magnitude of CD4bs-specific, including VRC01-class, B cells | Measured 2 weeks after the 3rd vaccination at week 28
  Measured by BCR sequencing of sorted B cells
Response rate of vaccine-specific and CD4bs-specific binding antibodies | Measured 6 months and 12 months after the 3rd vaccination at week 28
  Measured by BAMA
Magnitude of vaccine-specific and CD4bs-specific binding antibodies | Measured 6 months and 12 months after the 3rd vaccination at week 28
  Measured by BAMA
Response rate of CD4bs-specific memory B cells | Measured 6 months and 12 months after the 3rd vaccination at week 28
  Measured by flow cytometry
Response rate of serum neutralization | Measured 6 months and 12 months after the 3rd vaccination at week 28
  Measured by TZM-bl assay
Magnitude of serum neutralization | Measured 6 months and 12 months after the 3rd vaccination at week 28
  Measured by TZM-bl assay
EPI vaccine-specific binding antibody responses | Measured 2 weeks, 6 months, and 12 months after the 3rd vaccination at week 28
  Assessed by Pediatric Vaccine Multiplex Assay (PVMA)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Violari, Study Chair — Perinatal HIV Research Unit
Locations (1):
- Soweto HVTN CRS, Soweto, Gauteng, South Africa